CLINICAL TRIAL: NCT02297308
Title: A Single Center, Retrospective Study Evaluating the Use of the SoloPath® Sheath in Reducing Vascular and Bleeding Complications After Transcatheter Aortic Valve Implantation
Brief Title: A Retrospective Study Evaluating the Use of the SoloPath® Sheath in Reducing Vascular and Bleeding Complications
Status: Completed | Type: Observational
Sponsor: Terumo Medical Corporation (Industry)
Collaborators: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TIS2014-001
Record Dates: First submitted 2014-10-21; First posted 2014-11-21 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Vascular Access Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SoloPath Sheath: The study focuses on subjects that underwent TAVI with a SoloPath Sheath used for femoral vascualar access

SUMMARY:
This study is a retrospective, single center data collection to assess bleeding and vascular complications associated with TAVI when a SoloPath® Balloon Expandable TransFemoral Introducer is used for vascular access.

DETAILED DESCRIPTION:
This study is intended to collect data on the rate of vascular complications in subjects having transfemoral TAVI when the SoloPath® Balloon Expandable TransFemoral Introducer is used as a guide for introduction and delivery of TAVI devices. The use of a small profile sheath could possibly reduce the incidence of post procedure vascular complications associated with TAVI and further enhance the safety of accessing the femoral delivery route.

In addition, this study will examine the impact of arterial morphology and other subject risk factors as a predictor of clinical outcomes within 30 days following TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have undergone a TAVI procedure with femoral access achieved with a 19Fr (ID) SoloPath (STFI) sheath.
2. Male or female ≥ 18 years old.

Exclusion Criteria:

1. Subjects with Femoral or Iliac vessels less than 6mm on side of TAVI access will be excluded.
2. Subjects treated before January 1, 2011, are excluded from this analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects with severe aortic stenosis who underwent TAVI utilizing the SoloPath sheath for vascular access since 2011.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Asagr, M.D., Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between October 7th, 2014 and February 9th, 2015 at the Montreal Heart Institute.
Groups:
- SoloPath Sheath: The study focused on subjects that underwent TAVI with a SoloPath Sheath used for femoral vascular access.
Period: Overall Study
Arm/Group | SoloPath Sheath
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SoloPath Sheath
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 44
Region of Enrollment [Number; unit: participants]
  Canada | 90

OUTCOME MEASURES:

1. Primary Outcome: Vascular Access Site Complications
Description: Rate of VARC-2 defined vascular complications within 30 days of TAVI.
Time Frame: withn 30 days of TAVI procedure
Measure: Number; unit: participants
Groups:
- SoloPath Sheath: Vascular Complications
Arm/Group | SoloPath Sheath
Number analyzed (Participants) | 90
participants | 17

2. Secondary Outcome: Bleeding Complications at the Access Site
Description: VARC-2 defined vascular access site bleeding complications i.e. minor, major or life threatening bleeding
Time Frame: within 30 days of TAVI procedure
Measure: Number; unit: participants
Groups:
- SoloPath Sheath: Rate of VARC-2 defined access site bleeding complications.
Arm/Group | SoloPath Sheath
Number analyzed (Participants) | 90
participants | 19

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed as this was a retrospective study.
Arm/Group | SoloPath Sheath
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Single center, retrospective data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall be permitted to publish the results of the study in a manner that fairly and accurately sets forth the conclusions reached. The party seeking publication shall submit to the sponsor for review a draft of the proposed publication at least thirty (30) days prior to submission of the draft for publication.